CLINICAL TRIAL: NCT01783561
Title: Early Versus Routine Caffeine Administration in Extremely Preterm Neonates
Acronym: EARLYCAFFEINE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sharp HealthCare (Other)
Responsible Party: Principal Investigator, Anup Katheria, M.D., Director of Neonatal Research, Sharp HealthCare
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2HRCAFFEINE
Record Dates: First submitted 2013-01-31; First posted 2013-02-05 (Estimated); Results first posted 2017-08-01 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-11

CONDITIONS: Caffeine
Keywords: caffeine; intubation; hemodynamic
MeSH Terms: interventions — Caffeine; caffeine citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- early caffeine (Active Comparator): Infants will receive a blinded dose of either placebo (IV normal saline) or IV caffeine citrate 20mg/kg infused over 15 minutes within the first 2 hours of life. If the infant is in the early caffeine group, the blinded drug will be IV caffeine citrate 20mg/kg in the first 2 hours and placebo at 12 hours of life.
  Interventions: Drug: Caffeine
- Routine caffeine (Placebo Comparator): Infants will receive a blinded dose of either placebo (IV normal saline) or IV caffeine citrate 20mg/kg infused over 10 minutes within the first 2 hours of life. If the infant is in the routine caffeine group, the blinded drug will be placebo in the DR and IV caffeine citrate 20mg/kg at 12 hours of life.
  Interventions: Drug: Caffeine

INTERVENTIONS:
Drug: Caffeine — Infants will receive a blinded dose of either placebo (IV normal saline) or IV caffeine citrate 20mg/kg infused over 10 minutes within the first 2 hours of life. They will receive a blinded dose of the opposite of what they received in the DR (placebo or caffeine) at 6 hours of life. Therefore, the intervention is timing of initial caffeine dose.
  Other Names: caffeine citrate; IV caffeine

SUMMARY:
Premature infants are at risk of having pauses in breathing, or apneas, due to their immaturity. Premature infants are routinely given caffeine, a respiratory stimulant, on the first day of life to prevent apneas. However, if they continue to have apneas, they may require a breathing tube to be placed in the trachea. There are risks to having a breathing tube, so it would be beneficial to avoid it if possible. If caffeine is given earlier, it may decrease the need for a breathing tube. Some studies also suggest that caffeine may also improve heart function which may prevent low blood pressure if given early.

DETAILED DESCRIPTION:
This goal of this observational study is to compare the respiratory and acute hemodynamic effects of caffeine administered in the first 2 hours versus 12 hours of life in infants <29 weeks gestation. Our primary hypothesis is that caffeine administered in the first two hours of life can prevent the need for endotracheal intubation in the first 12 hours of life.. These evaluations are critical in determining both the safety and efficacy of early caffeine therapy.

ELIGIBILITY:
Inclusion Criteria:

* Any infant delivered at Sharp Mary Birch Hospital between 23 and 28 6/7 weeks; gestation

Exclusion Criteria:

* Any infant with a major congenital anomaly including airway anomalies, congenital diaphragmatic hernia, or hydrops
* Any infant with a known or a discovered major cardiac defect other than a patent ductus arterious (PDA), patent foramen ovale (PFO), or small ventricular septal defect (VSD)
* Inability to place a peripheral IV after two attempts. Severe apnea or bradycardia in the first 60 minutes of life requiring emergent endotracheal intubation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anup Katheria, MD, Principal Investigator — Sharp HealthCare
Locations (1):
- Sharp Memorial Hospital, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Early Caffeine: Infants will receive a blinded dose of either placebo (IV normal saline) or IV caffeine citrate 20mg/kg infused over 15 minutes within the first 2 hours of life. If the infant is in the early caffeine group, the blinded drug will be IV caffeine citrate 20mg/kg in the first 2 hours and placebo at 12 hours of life.
  Caffeine: Infants will receive a blinded dose of either placebo (IV normal saline) or IV caffeine citrate 20mg/kg infused over 10 minutes within the first 30 minutes of life. They will receive a blinded dose of the opposite of what they received in the DR (placebo or caffeine) at 6 hours of life. Therefore, the intervention is timing of initial caffeine dose.
- Routine Caffeine: Infants will receive a blinded dose of either placebo (IV normal saline) or IV caffeine citrate 20mg/kg infused over 10 minutes within the first 2 hours of life. If the infant is in the routine caffeine group, the blinded drug will be placebo in the DR and IV caffeine citrate 20mg/kg at 12 hours of life.
  Caffeine: Infants will receive a blinded dose of either placebo (IV normal saline) or IV caffeine citrate 20mg/kg infused over 10 minutes within the first 30 minutes of life. They will receive a blinded dose of the opposite of what they received in the DR (placebo or caffeine) at 6 hours of life. Therefore, the intervention is timing of initial caffeine dose.
Period: Overall Study
Arm/Group | Early Caffeine | Routine Caffeine
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Caffeine | Routine Caffeine | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 10 | 21
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Intubation
Description: The primary aim of our study is to compare the respiratory effects of caffeine administered in the first 2 hours versus at 12 hours of life in infants <29 weeks' gestation. Our primary hypothesis is that early caffeine administered (at < 2 hours of life) can prevent the need for endotracheal intubation in the first 12 hours of life.
Time Frame: First 12 hours of life
Measure: Number; unit: participants
Arm/Group | Early Caffeine | Routine Caffeine
Number analyzed (Participants) | 11 | 10
participants | 3 | 7

2. Secondary Outcome: Subjects Requiring Inotropes in the First 24 Hours
Description: To determine if a loading dose of intravenous caffeine administered to preterm infants (< 29 weeks) within the first 2 hours of life compared to 12 hours of life decreases the need for inotropes for hypotension within the first 24 hours of life.
Time Frame: first 24 hours of life
Measure: Count of Participants; unit: Participants
Arm/Group | Early Caffeine | Routine Caffeine
Number analyzed (Participants) | 11 | 10
Participants | 0 | 2

3. Secondary Outcome: Systemic Blood Flow
Description: To determine if a loading dose of intravenous caffeine administered to preterm infants (< 29 weeks) within the first 2 hours of life compared to 12 hours of life results in improved measures of systemic blood flow (measured by superior vena cava flow)
Time Frame: first 24 hours
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Early Caffeine | Routine Caffeine
Number analyzed (Participants) | 11 | 10
ml/kg/min
  SVC flow | 101 (25) | 77 (24)
  RVO | 273 (62) | 219 (43)

ADVERSE EVENTS:
Arm/Group | Early Caffeine | Routine Caffeine
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No